CLINICAL TRIAL: NCT06014320
Title: Understanding the Alterations in Coagulation Factor Levels in Patients With End Stage Liver Disease
Brief Title: Alterations in Coagulation Factor Levels in Patients With End Stage Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexandra Ruan, Clinical Assistant Professor, Stanford University
Other Study IDs: 71275
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Liver Cirrhosis; Hemophilia; Hemophilia A; Hemophilia B; Liver Transplant Disorder; Liver Failure; Coagulation Factor Deficiency
Keywords: liver transplant; hemophilia; coagulation; thrombosis; bleeding; cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hemophilia A; Hemophilia B; Liver Failure; Thrombosis; Hemorrhage; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESLD: All participants recruited will belong to this group. These participants will all have end stage liver disease and be listed for liver transplant with an accepted organ offer.

SUMMARY:
The goal of this observational study is to learn about the changes in coagulation factor VIII and IX levels in patients undergoing liver transplantation to help guide future management of coagulation factor replacement in patients with hemophilia and liver disease. The question we aim to answer is: should the recommendations for factor replacement in patients with hereditary bleeding disorders be altered in the setting of end stage liver cirrhosis?

Participants will be asked to provide two blood samples, one at the beginning of their liver transplant, and one after their liver transplant.

DETAILED DESCRIPTION:
Current guidelines for management of hemophilia B suggest replacement of factor IX to 100% prior to major abdominal surgery. However, in patients with concurrent liver cirrhosis where the liver does not produce Factor IX, is it worth considering adjusting the factor replacement strategy? We recently had a case of a patient with Hemophilia B and end-stage liver disease (ESLD) who underwent orthotopic liver transplantation and received the standard pre-operative recombinant factor IX replacement. His case was complicated by intra-cardiac thrombus and hypotension. We conduct a small study to assess the pre-operative thromboelastography (TEG) and factor levels in ESLD patient which we hope will help guide clinical decision making in future hemophilia B patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* participants who have end stage liver disease who are listed for liver transplantation and have an accepted organ offer
* age > 18+
* MELD > 25

Exclusion Criteria:

* undergoing multi-organ transplant
* tumor MELD exception points
* has hereditary coagulation disease
* currently on therapeutic blood thinner or anti-platelet medication (ie. aspirin, plavix, warfarin, heparin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited for the study who have end stage liver disease and are undergoing liver transplant at Stanford hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Factor VIII level | 12 hours
  We will collect Factor VIII level pre- and post- transplant
Factor IX level | 12 hours
  We will collect Factor IX level pre- and post- transplant
Thromboelastography (TEG) values | 12 hours
  We will collect thromboelastography values pre- and post- transplant

SECONDARY OUTCOMES:
Complications | 24 hours
  We will collect data on bleeding or clotting events during the liver transplant surgery and 24 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Ruan, MD, Study Director — Stanford University; Martin Angst, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso Madrigal C, Dobon Rebollo M, Laredo de la Torre V, Palomera Bernal L, Garcia Gil FA. Liver transplantation in hemophilia A and von Willebrand disease type 3: perioperative management and post-transplant outcome. Rev Esp Enferm Dig. 2018 Aug;110(8):522-526. doi: 10.17235/reed.2018.5204/2017. PMID 29931985
- [Background] Togashi J, Akamatsu N, Tanaka T, Sugawara Y, Tsukada K, Kaneko J, Arita J, Sakamoto Y, Hasegawa K, Kokudo N. Living donor liver transplantation for hemophilia with special reference to the management of perioperative clotting factor replacement. Liver Transpl. 2016 Mar;22(3):366-70. doi: 10.1002/lt.24341. Epub 2016 Feb 15. No abstract available. PMID 26390184
- [Background] Kadry Z, de Moerloose P, Giostra E, Morel P, Huber O, Meili E, Blum HE, Mentha G. Orthotopic liver transplantation in hemophilia B: a case report. Transpl Int. 1995;8(6):485-7. doi: 10.1007/BF00335602. PMID 8579741
- [Result] Ramiz S, Hartmann J, Young G, Escobar MA, Chitlur M. Clinical utility of viscoelastic testing (TEG and ROTEM analyzers) in the management of old and new therapies for hemophilia. Am J Hematol. 2019 Feb;94(2):249-256. doi: 10.1002/ajh.25319. Epub 2018 Dec 7. PMID 30328141